CLINICAL TRIAL: NCT01380665
Title: Prospective, Single Arm, Post-Marketing Trial to Examine the Safety and Functionality of the Prevena™ Incision Management System, A Negative Pressure Based Surgical Wound Management System, Over Primarily Closed Hip and Knee Incisions in Patients Immediately Post Total Hip and Knee Arthroplasty
Brief Title: Prevena™ Incision Management System Over Primarily Closed Hip and Knee Incisions in Patients Immediately Post Total Hip and Knee Arthroplasty
Acronym: Prevena2009-45
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: KCI USA, Inc (Industry)
Responsible Party: Sponsor
Organization: Solventum US LLC (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Prevena2009-45
Record Dates: First submitted 2011-06-09; First posted 2011-06-27 (Estimated); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Linear or Emi-linear Incisions; Total Hip Arthroplasty; Total Knee Arthroplasty
Keywords: Prevena; Incision; Management; System; total; knee; hip; replacement; Surgery; Negative; Pressure; dressing; KCI
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- There is one group of 100 patients (Other): 50 of these patients will receive a total hip replacement; 50 patients will receive a total knee replacement;
  Interventions: Device: Prevena Incisional Management System

INTERVENTIONS:
Device: Prevena Incisional Management System — All evaluable patients will utilize the Prevena Incisional Management System

SUMMARY:
The intent of this study is to evaluate the Prevena ™ 125 Unit and dressing system, when applied to either the hip or knee area over a surgical cut for the time you are hospitalized.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be ≥ 18 years of age
2. Subject must, at the treating physician's determination and definition, be an appropriate Candidate for primary total hip or knee arthroplasty
3. Subjects who undergo primary total knee or hip arthroplasty must have a linear or semi-linear incision whose length and curvature should fit within the dimensions bound by the polyurethane foam (10 inches in length by 2.5 inches in width)
4. Subject is able and willing to provide written informed consent and comply with visit schedule
5. Subject must agree to avoid application of tanning lotions or exposure of ultraviolet radiation from sun or artificial sources such as a tanning bed on operative area for the duration of study participation
6. Subject must not be pregnant if of child-bearing potential, or otherwise must be surgically sterilized or unable to conceive. All females, regardless of child-bearing potential, will receive a urine hCG test 2 weeks prior to surgery and the test result must be negative for pregnancy.
7. Subjects who are of child-bearing potential must be utilizing an acceptable method of birth control (eg, birth control pills, condom with spermicide, diaphragm with spermicide, implants, IUD, injections, vaginal rings, hormonal skin patch, etc) and be willing to continue birth control for duration of study participation. If birth control method is the form of birth control pills, shots, implants skin patches, or IUD, the method must have been utilized for at least 30 days prior to study participation.
8. Subject must be willing to wear loose fitting clothing for duration of treatment period
9. Subject must be willing to comply with visit schedule for the duration of the study

Exclusion Criteria:

1. Positive pregnancy test confirmed by hCG in urine
2. Current or past (30 days prior to surgery) within time of screening attempts to become pregnant
3. Current local or systemic infection (eg, skin infections, sinus infections, urinary tract infection, sepsis, etc)
4. Current or past (14 days prior to surgery) within time of screening topical treatments on operative area (eg, laser hair or tattoo removal, sunless tanning lotions)
5. Current or past (14 days prior to surgery) steroid topical therapies on operative area
6. Current or past (30 days prior to surgery) use of oral steroids (NOTE: Use of non-topical, ophthalmic or aerosol types of steroids (ie, inhaled corticosteroids) are permitted at screening and throughout the clinical trial)
7. Current or past (72 hours prior to surgery) within surgery use of antihistamines
8. Current or past (30 days prior to surgery) within time of screening use of oral Tetracycline or AcutaneTM or topical Tetracycline or AcutaneTM on the operative area
9. Presence of skin lesions or abnormalities on operative area
10. Current or past malignancy requiring immunosuppressant therapy or chemotherapy within 5 years within time of screening
11. Presence of excessive skin folds on operative area
12. Intentional exposure of the operative area to ultraviolet radiation (14 days prior to surgery) within time of screening (ie, sunbathing or tanning bed)
13. Presence of sunburned or peeling skin on operative area
14. Tattoos on operative area
15. Presence of severe, raised scar tissue on operative area which may interfere with pre and post skin evaluation assessments
16. Presence of an open wound prior to the index surgical procedure on operative area
17. Reported alcohol (≥ 3 drinks per day) or drug abuse within the past 6 months
18. Topical hypersensitivity or allergy to any disposable components of the dressing system (eg, silver, polyurethane, polyester, or acrylic adhesive)
19. Topical hypersensitivity or allergy towards any medical adhesive
20. Current enrollment or past participation in this clinical study or any other study within ≤30 days
21. Any systemic or local active dermatological disease that might interfere with the evaluation of the operative area (eg, Meleney's ulcer, scleroderma, chronic urticaria, psoriasis, skin cancer, eczema, seborrhea, or malignancy)
22. Connective tissue disease or collagen vascular disease (eg, Ehlers-Danlos syndrome, systemic lupus erythematosus, rheumatoid arthritis)
23. Current or history of hematological disorders or conditions (eg, polycythemia vera, thrombocythemia, sickle-cell disease)
24. Any Subject with conditions which can potentially result in abnormally pigmented skin (eg, melasma, vitiligo, pityriasis versicolor)
25. Inability or refusal to wear loose fitting clothing for the duration of the treatment period
26. Subjects in whom orthopaedic reconstruction is required in addition to total hip or knee arthroplasty
27. Subjects who are having the total hip or knee arthroplasty as a result of acute orthopaedic trauma
28. Subjects who have incurred acute orthopaedic trauma (ie, hip fracture) recently or at any time
29. Subjects who have either acute or chronic open/active wounds present (including biopsies, ulcerations, etc)
30. Subjects in whom the index procedure is a revision of a total hip or knee arthroplasty
31. Subjects in whom the primary or partial total hip or knee arthroplasty would also be performed on the contra lateral knee or hip at the same time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Negative pressure environment with accurate and reliable indicators;Dressing biocompatible with incision site and skin;Minimal dressing changes during therapy;Acceptable safety profile; minimal/no AEs;Patient comfort and dressing integrity after surgery | during hospitalization (up to 7 days) and thru follow-up 30 days after dressing removal